CLINICAL TRIAL: NCT03112928
Title: Phantom Motor Execution Via Myoelectric Pattern Recognition, Virtual and Augmented Reality, and Serious Gaming as a Treatment of Phantom Limb Pain
Brief Title: Phantom Motor Execution Via MPR, VR/AR, and SG, as a Treatment of PLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrum (Industry)
Collaborators: Chalmers University of Technology (Other); Sahlgrenska University Hospital (Other); Örebro University, Sweden (Other); Bräcke Diakoni, Sweden (Unknown); University Rehabilitation Institute, Republic of Slovenia (Other); University Medical Center Groningen (Other); University of New Brunswick (Other); National University of Ireland, Galway, Ireland (Other); Shirley Ryan AbilityLab (Other); Ruhr University of Bochum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 007733
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2020-09

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: International, multi-centre, double-blind, randomized, controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be informed that both treatments have been shown effective in previous studies, and in the present study we are comparing their efficacy.
  The person conducting the pain evaluation (outcomes assessor) will not treat the participants and will be unaware of which treatment is given to each participant. The person treating the subject is different than the person evaluating.
  The principal and coordinating investigator will receive blinded data from all participating centers to analyze the clinical trial outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phantom Motor Execution (PME) (Experimental): Phantom motor execution is decoded via myoelectric pattern recognition and promoted via serious gaming in virtual and augmented reality.
  Interventions: Device: Phantom Motor Execution
- Phantom Motor Imagery (PMI) (Active Comparator): Use the same device and visual stimulation as PME, with the difference that participants imagine to perform, rather than execute phantom movements. Myoelectric activity is used to monitor that the subjects do not produce muscular contractions but only imagine the movements.
  Interventions: Device: Phantom Motor Imagery

INTERVENTIONS:
Device: Phantom Motor Execution — Neuromotus - PME decodes motor volition applying machine learning to surface electromyography. Once the intention of movement is known, this is use to control serious games in virtual and augmented reality.
  A treatment session of MPE consists of:
  1. Pain evaluation
  2. Placement of the electrodes and fiducial marker
  3. Practice of motor execution in Augmented Reality (AR)
  4. Gaming using phantom movements
  5. Practice of motor execution by matching random target postures of a virtual limb.
  Step 3 to 4 are repeated for different phantom joints, initially one at the time progressing to several joints simultaneously. A treatment session last 2 hours.
  Other Names: Neuromotus - PME
  Arms: Phantom Motor Execution (PME)
Device: Phantom Motor Imagery — The only difference between PME and PMI is that in the former myoelectric signals are used to give the participants control over the virtual environments, whereas in PMI the presence of myoelectric activity is used as an alarm to remind the participant that it must imagine rather than execute the phantom movement. In PMI the virtual environments act autonomously to guide the participant in imagination of movement.
  Other Names: Neuromotus - PMI
  Arms: Phantom Motor Imagery (PMI)

SUMMARY:
This international, multi-center, double-blind, randomized, controlled clinical trial aims to evaluate the efficacy of Phantom Motor Execution (PME) and Phantom Motor Imagery (PMI) as treatments of Phantom Limb Pain (PLP). In PME, myoelectric pattern recognition (MPR) is used to predict motor volition and then use the decoded movements to control virtual and augmented reality environments (VR/AR), along with serious gaming (SG). The same device and VR/AR environments are used in PMI with the difference that subjects will imagine rather than execute phantom movements. Electromyography is used to monitor for no muscular activity in PMI.

DETAILED DESCRIPTION:
Sixty-six subjects with upper or lower limb amputations are planned to take part in this study. Subjects will be assigned randomly to PME and PMI treatments (2:1 proportion). After treatment completion (15 sessions of 2 hours each) and follow-up period of six months, patients that received PMI will be given the choice to receive PME. The design is double blinded as the patient will be informed that the treatment received, regardless of which, has been shown effective in previous studies. The person conducting the pain evaluations will be blinded to which treatment each patient receives, and will not take part on providing treatment (evaluator and therapist are different persons).

ELIGIBILITY:
* Subject must be older than 18 years.
* If the subjects are under pharmacological treatments, there must be no variations on the medicament dosages for at least one month (steady consumption).
* The last session of previous treatments must be at least 3 months old.
* Any pain reduction potentially attributed to previous phantom limb pain treatments must be at least 3 months old.
* Subjects must have control over at least a portion of biceps and triceps muscles for upper limb amputations, and quadriceps and hamstrings for the lower limb amputations.
* The subject has signed a written informed consent.
* The subject must be in a stable prosthetic situation (i.e. satisfied with the fitting of the prosthesis) or being a non user.
* At least six months should be passed since the amputation: acute phantom limb pain cases should not be included in the study.
* The patient subject should not have a significant cognitive impairment that prevents the patient from following instructions.
* Subjects with abundant soft tissue on their stump will not be automatically excluded, however, an evaluation in the system is required to analyze if sufficient electromyography signals can be recorded.
* Subjects for whom skin contact or muscle contraction are painful (NRS > 2) are not eligible for the study.
* The subject should not have any condition associated with risk of poor protocol compliance.
* The subject should not have any other condition or symptoms preventing the patient from entering the study, according to the investigator´s judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Pain Rating Index registered at the beginning (1st session) and at the end of the treatment (15th session). | 28-40 weeks, depending on the frequency of the sessions.
  The Pain Rating Index (PRI) is calculated as the sum of 15 descriptors. At the end of each treatment session the descriptors are presented to the patient, who rates each of them with an intensity scale from 0 to 3. The PRI is therefore a number between 0 and 45: the higher the index the greater is the pain. The primary efficacy variable for this study is the change in PRI between the first and the last treatment session.

SECONDARY OUTCOMES:
Pain Disability Index registered at the beginning (1st session) and the end of the treatment (15th session). | 28-40 weeks, depending on the frequency of the sessions.
  The Pain Disability Index (PDI) measures the impact that pain has on the ability of a person to participate in essential life activities. The index is comprised between 0 and 70. The higher the index the greater the person's disability due to pain is. The secondary efficacy variable of this study is the change in PDI between the first and the last treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Max Ortiz Catalan, PhD, Principal Investigator — Chalmers Technological University
Locations (9):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States
- Institue of Biomedical Engineering, University of New Brunswick, Fredericton, New Brunswick, Canada
- Department of Psychosomatic Medicine and Psychotherapy, LWL University Hospital, Ruhr - University Bochum (RUB), Bochum, Germany
- School of Psychology, National University of Ireland, Galway, Connacht, Ireland
- University of Groningen, University Medical Center Groningen, Department of Rehabilitation Medicine, Groningen, Netherlands
- University Rehabilitation Institute, Ljubljana, Slovenia
- Sweden (3):
  - Ortopedteknik, Region Örebro län, Örebro, Närke
  - Bräcke Diakoni, Stockholm, Uppland
  - Gåskolan, Ortopedtekniska avdelningen, Gothenburg, Västergötland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortiz-Catalan M, Guethmundsdottir RA, Kristoffersen MB, Zepeda-Echavarria A, Caine-Winterberger K, Kulbacka-Ortiz K, Widehammar C, Eriksson K, Stockselius A, Ragno C, Pihlar Z, Burger H, Hermansson L. Phantom motor execution facilitated by machine learning and augmented reality as treatment for phantom limb pain: a single group, clinical trial in patients with chronic intractable phantom limb pain. Lancet. 2016 Dec 10;388(10062):2885-2894. doi: 10.1016/S0140-6736(16)31598-7. Epub 2016 Dec 2. PMID 27916234
- [Background] Ortiz-Catalan M, Sander N, Kristoffersen MB, Hakansson B, Branemark R. Treatment of phantom limb pain (PLP) based on augmented reality and gaming controlled by myoelectric pattern recognition: a case study of a chronic PLP patient. Front Neurosci. 2014 Feb 25;8:24. doi: 10.3389/fnins.2014.00024. eCollection 2014. PMID 24616655
- [Derived] Lendaro E, Van der Sluis CK, Hermansson L, Bunketorp-Kall L, Burger H, Keesom E, Widehammar C, Munoz-Novoa M, McGuire BE, O'Reilly P, Earley EJ, Iqbal S, Kristoffersen MB, Stockselius A, Gudmundson L, Hill W, Diers M, Turner KL, Weiss T, Ortiz-Catalan M. Extended reality used in the treatment of phantom limb pain: a multicenter, double-blind, randomized controlled trial. Pain. 2025 Mar 1;166(3):571-586. doi: 10.1097/j.pain.0000000000003384. Epub 2024 Sep 5. PMID 39250328
- [Derived] Lendaro E, Earley EJ, Ortiz-Catalan M. Statistical analysis plan for an international, double-blind, randomized controlled clinical trial on the use of phantom motor execution as a treatment for phantom limb pain. Trials. 2022 Feb 13;23(1):138. doi: 10.1186/s13063-021-05962-7. PMID 35152915
- [Derived] Lendaro E, Hermansson L, Burger H, Van der Sluis CK, McGuire BE, Pilch M, Bunketorp-Kall L, Kulbacka-Ortiz K, Rigner I, Stockselius A, Gudmundson L, Widehammar C, Hill W, Geers S, Ortiz-Catalan M. Phantom motor execution as a treatment for phantom limb pain: protocol of an international, double-blind, randomised controlled clinical trial. BMJ Open. 2018 Jul 16;8(7):e021039. doi: 10.1136/bmjopen-2017-021039. PMID 30012784